CLINICAL TRIAL: NCT01534780
Title: A Controlled Randomized Study of Protack, Securestrap and Glubran Glue as Fixation Devices in Laparoscopic Ventral Herniotomy
Brief Title: 3 Fixation Devices in Laparoscopic Ventral Herniotomy
Acronym: FS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Horsens Hospital (Other)
Collaborators: Randers Regional Hospital (Other)
Responsible Party: Principal Investigator, Hans Friis-Andersen, Principal Investigator, Horsens Hospital
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: KIR-001-HRH
Record Dates: First submitted 2012-02-09; First posted 2012-02-17 (Estimated); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Ventral Hernia
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- fixation with Protack (Experimental)
  Interventions: Procedure: laparoscopic ventral herniotomy; Device: Protack
- fixation with Securestrap (Experimental)
  Interventions: Procedure: laparoscopic ventral herniotomy; Device: Securestrap
- fixation with Glubran (Experimental): surgery
  Interventions: Procedure: laparoscopic ventral herniotomy; Device: Glubran

INTERVENTIONS:
Procedure: laparoscopic ventral herniotomy — Laparoscopy in general anesthesia are performed with placement of Physiomesh intraperitoneally. Fixation of the mesh is performed with 1 of 3 possible devices
  Other Names: no other names
Device: Protack — fixation of mesh with protack
  Arms: fixation with Protack
Device: Securestrap — fixation of mesh with Securestrap
  Arms: fixation with Securestrap
Device: Glubran — fixation of mesh with Glubran
  Arms: fixation with Glubran

SUMMARY:
Clinical, controlled, randomized, prospective study. Ventral hernias between 2(1.5)cm and 7 cm, laparoscopic surgery with intraperitoneal onlay mesh.

Three randomization groups of 25 patients giving a total of 75 patients. Mesh is fixated with either Protack, Securestrap or Glubran II. Primary outcome: postoperative pain on the 2nd postoperative day. Secondary outcomes: pain, quality of life, recurrence and adhesions at 1, 6, 12, 24, 36, 48 and 60 months postoperative.

DETAILED DESCRIPTION:
see brief summary

ELIGIBILITY:
Inclusion Criteria:

* ventral hernia 2(1,5) < dia > 7 cm
* danish speaking
* of sound mind
* bmi < 35
* ASA 3 or less, no contra indication against laparoscopy

Exclusion Criteria:

* other size hernias,
* no danish,
* bmi > 35

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2013-04; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Pain | 1 measurement, 2nd postoperative day
  Dolo Test (VAS)

SECONDARY OUTCOMES:
hernia recurrence | 7 measurements, postoperative month 1, 6, 12, 24, 36, 48 and 60
  clinical examination and perhaps CT scan
quality of life | 7 measurements, postoperative month 1, 6, 12, 24, 36, 48 and 60
  SF 36 and Carolina's Comfort Scale
Pain | 7 measurements, day 1, 3 and 4 and postoperative month 1, 6, 12, 24
  Dolo Test(VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Sanne S Harsløf, MD, Study Chair — Regionshospitalet Horsens; Thorbjørn Sommer, MD, PhD, Study Director — Randers Regional Hospital
Locations (1):
- Regional Hospital Horsens, Horsens, Denmark

REFERENCES:
- [Derived] Harslof S, Krum-Moller P, Sommer T, Zinther N, Wara P, Friis-Andersen H. Effect of fixation devices on postoperative pain after laparoscopic ventral hernia repair: a randomized clinical trial of permanent tacks, absorbable tacks, and synthetic glue. Langenbecks Arch Surg. 2018 Jun;403(4):529-537. doi: 10.1007/s00423-018-1676-z. Epub 2018 May 25. PMID 29799075